CLINICAL TRIAL: NCT04322851
Title: Implication of B-line Estimated by Lung Ultrasound on Risk of Reintubation in Mechanically Ventilated Patients With Acute Decompensated Heart Failure
Brief Title: B-line by Lung US in Patients With Acute Decompensated Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Min-Seok Kim, professor of medicine, Asan Medical Center
Other Study IDs: AMC_2020_0164
Record Dates: First submitted 2020-02-26; First posted 2020-03-26 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- B-line positive
  Interventions: Diagnostic Test: Lung ultrasound
- B-line negative
  Interventions: Diagnostic Test: Lung ultrasound

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Lung ultrasound performed at the time of extubation to evaluate B-line in patients with mechanical ventilation due to acute decompensated heart failure

SUMMARY:
The purpose of this study is to evaluate that B-line detected by lung ultrasound before extubation in patients with acute decompensated heart failure can predict future risk of reintubation and clinical outcomes during admission in Korea.

ELIGIBILITY:
Inclusion Criteria:

* mechanical ventilation due to acute heart failure

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who are on mechanical ventilation due to acute heart failure
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Re-intubation rate | within 72 hours from initial extubation

CONTACTS AND LOCATIONS:
Overall Officials: Minseok Kim, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided